CLINICAL TRIAL: NCT06431763
Title: A Randomized, Multicenter, Open-label Trial Comparing the Effectiveness of Inclisiran to Bempedoic Acid on LDL Cholesterol (LDL-C) Lowering in Participants With Atherosclerotic Cardiovascular Disease (VICTORION-CHALLENGE)
Brief Title: A Study to Investigate LDL-cholesterol Lowering With Inclisiran Compared to Bempedoic Acid in Patients With Atherosclerotic Cardiovascular Disease.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CKJX839A1DE02
Record Dates: First submitted 2024-04-30; First posted 2024-05-29 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Hypercholesterolemia
Keywords: LDL-cholesterol; atherosclerotic cardiovascular disease; Inclisiran; bempedoic acid; BPA; PCSK9 inhibitor; head-to-head comparison
MeSH Terms: conditions — Hypercholesterolemia; Atherosclerosis | interventions — RNA, Small Interfering

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inclisiran (Experimental): Inclisiran treatment on top of background treatment (high intensity statin with/without ezetimibe)
  Interventions: Drug: Inclisiran sodium
- Bempedoic acid (BPA) (Active Comparator): BPA treatment on top of background treatment (high intensity statin with/without ezetimibe)
  Interventions: Drug: BPA

INTERVENTIONS:
Drug: Inclisiran sodium — 300 mg s.c. administered at day 1 and day 90
  Other Names: PCSK9 inhibitor, siRNA
  Arms: Inclisiran
Drug: BPA — 180 mg daily per oral
  Other Names: small molecule, ACL inhibitor
  Arms: Bempedoic acid (BPA)

SUMMARY:
This study is a phase IV, open-label, randomized study designed to evaluate the efficacy of Inclisiran vs. bempedoic acid (BPA) in 400 adult subjects (≥ 18 years) at very high and high risk for cardiovascular events as defined by the cardiovascular risk categories in the 2019 ESC/EAS guidelines for the management of dyslipidemias (Mach et al 2020) and elevated levels of LDL-C (≥ 70 mg/dL) despite being on a maximally tolerated high-intensity (HI) statin dose (+/- Ezetimibe). Currently, BPA is recommended ahead of injectables by German HTA body (GBA). A head-to-head trial is proposed to provide robust scientific data on the superiority of Inclisiran vs. BPA and to support the early use of Inclisiran.

DETAILED DESCRIPTION:
During the screening period study eligibility will be assessed and the participants' individual LDL-C target according to guideline (Mach et al., 2020) will be determined. Among other criteria, at screening, a participant must be on a stable maximally tolerated dose of a HI statin with either atorvastatin ≥40 mg once a day (QD) or rosuvastatin ≥20 mg QD (+/- Ezetimibe [10mg]) for ≥ 4 weeks with which, however, a target LDL-C of < 70 mg/dL is not reached.

During the open-label treatment period, all participants, who fulfill the inclusion/exclusion criteria, will be randomized at V1 (Day 1) in a 1:1 open-label fashion to either Inclisiran sodium 300 mg s.c. (administered at Day 1 and Day 90) or to BPA tablets 180 mg p.o. (given once daily). Participants will be required to maintain their background lipid-lowering treatment (maximally tolerated statin dose +/- Ezetimibe) unchanged for the duration of the study. The end of treatment (EOT) is reached at day 150.

A Safety-Follow-up call will be conducted 30 days after EOT visit (Day 180).

The overall study duration is approximately 190 days but can vary depending on individual screening and the visit windows allowed for the treatment period and EOS visit.

ELIGIBILITY:
Inclusion Criteria:

1. Fasting LDL-C ≥ 70 mg/dL at screening
2. Participants must be on a stable (≥ 4 weeks) and well-tolerated lipid-lowering regimen (with or without Ezetimibe [10mg]) that must include a high-intensity statin therapy with either atorvastatin ≥40 mg QD or rosuvastatin ≥20 mg QD in a maximally tolerated or maximally approved dose at screening
3. Participants categorized as very high or high CV risk, as defined below:

   * Very high risk participants with at least one of the following:

     * Documented ASCVD: ACS: Unstable angina or myocardial infarction, Stable angina, Coronary revascularization, Unequivocally documented ASCVD upon prior imaging, Stroke and Transient Ischaemic Attack (TIA), Peripheral artery disease (PAD)
     * Diabetes mellitus (DM) with target organ damage (defined as microalbuminuria, retinopathy, or neuropathy), or at least ≥ 3 major risk factors, or early onset of Type 1 DM of long duration (< 20 years)
     * A calculated SCORE2 ≥ 7.5 % for age < 50 years; SCORE2 ≥ 10 % for age 50-69 years; SCORE2-OP ≥ 15 % for age ≥ 70 years to estimate 10-year risk of fatal and non-fatal CVD
     * Pre-existing diagnosis of heterozygous familial hyper-cholesterolemia (HeFH) with ASCVD or with another major risk factor OR
   * High risk participants with at least one of the following:

     * Markedly elevated single risk factors, in particular total cholesterol > 310 mg/dL, LDL-C > 190 mg/dL, or blood pressure ≥ 180/110 mmHg
     * Pre-existing diagnosis of HeFH without other major risk factors
     * DM without target organ damage (defined as microalbuminuria, retinopathy, or neuropathy), with DM duration ≥ 10 years or other additional risk factor
     * Moderate chronic kidney disease (eGFR 30-59 mL/min/1.73m2)
     * A calculated SCORE2 2.5 to < 7.5 % for age < 50 years; SCORE2 5 to < 10 % for age 50-69 years; SCORE2-OP 7.5 to < 15 % for age ≥ 70 years to estimate 10-year risk of fatal and non-fatal CVD as defined by the cardiovascular risk categories in the 2019 ESC/EAS guideline (Mach et al 2020), and updated SCORE2 and SCORE2-OP (Hageman et al 2021, de Vries et al 2021, Visseren et al 2021). Further details for documented ASCVD will be provided in the protocol.
4. Fasting triglyceride < 400 mg/dL at screening

Exclusion Criteria:

1. Acute coronary syndrome, ischemic stroke, peripheral arterial revascularization procedure or amputation due to atherosclerotic disease < 4 months prior to screening visit or V1.
2. Planned or expected cardiac, cerebrovascular or peripheral artery surgery or coronary re-vascularization within 6 months after screening visit.
3. Heart failure NYHA class IV at screening or V1.
4. Participants on more than one other lipid-lowering drug on top of statin at screening visit.
5. Previous treatment with a mAb directed towards PCSK9 (e.g., evolocumab, alirocumab) or planned use after screening visit.
6. Previous treatment prior to screening with BPA within 90 days
7. Previous exposure to Inclisiran or any other non-mAb PCSK9-targeted therapy, either as an investigational or marketed drug.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2024-06-21 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2026-01-02 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in LDL-C levels | Baseline, Day 150
  To demonstrate superiority of Inclisiran compared to BPA, in combination with standard of care (maximally tolerated HI statin dose +/- Ezetimibe) in reducing relative LDL-C levels at Day 150.

SECONDARY OUTCOMES:
Percent change from baseline in LDL-C levels in patients without Ezetimibe | Baseline, Day 150
  To demonstrate superiority of Inclisiran compared to BPA, in patients on maximally tolerated HI statin dose without Ezetimibe in relative reduction of LDL-C levels at Day 150.
Percent change from baseline in LDL-C levels in patients with Ezetimibe | Baseline, Day 150
  To demonstrate superiority of Inclisiran compared to BPA, in patients on maximally tolerated HI statin dose with Ezetimibe in reducing relative LDL-C levels at Day 150.
Number of participants by individual responsiveness | Day 150
  Number of patients who qualify for 'sufficient response' based on their individual risk class, defined through on treatment LDL-C levels.
  For patients classified as 'very high risk', responsiveness is 'achieved' once the LDL-C drops below 55mg/dL, and for patients classified as 'high risk' responsiveness is 'achieved' once the LDL-C < 70 mg/dL at Day 150.
Absolute change from Baseline in LDL-C | Day 150
  Assess efficacy of Inclisiran compared to BPA in reducing LDL-C (absolute reduction).
Percent change from Baseline in LDL-C levels | Baseline, from Day 30 up to Day 150
  Assess efficacy of Inclisiran compared to BPA in reducing LDL-C [time-adjusted percent change] starting Day 30 and up to Day 150.
Percent change from Baseline in LDL-C levels | Between Day 90 and Day 150
  Assess efficacy of Inclisiran compared to BPA in reducing LDL-C [time-adjusted percent change] between Day 90 and Day 150.
Mean change from baseline in MMAS-8 over time | From Baseline up to Day 150
  Assess adherence to lipid-lowering therapy over time in participants receiving Inclisiran compared to BPA on top of maximally tolerated HI statins (+/- Ezetimibe) using the Morisky 8-Item Medication Adherence Scale (MMAS-8).
  The Morisky Medication Adherence Scale is an assessment tool used to measure non-adherence in patient populations. It consists of seven yes/no questions and one 5-point Likert scale with a sum score ranging between 0 and 8 points. The higher score indicates higher adherence.
Mean change from Baseline in TSQM over time | From Baseline up to Day 150
  Assess effect of Inclisiran compared to BPA regarding treatment satisfaction using the Treatment Satisfaction Questionnaire for Medication (TSQM v. II).
  The TSQM (version II) comprises 11 items across four domains focusing on effectiveness (two items), side effects (four items), convenience (three items), and global satisfaction (two item) of the medication over the previous weeks, or since the patient's last use. With the exception of item 3 (presence of side effects; yes or no), all items have five or seven responses, scored from one (least satisfied) to five or seven (most satisfied). The 7-item scales had a nonneutral midpoint, such that there were more positive response options than negative response options, to allow for precise information to be obtained at the upper end of the score distribution. Item scores are summed to give four domain scores, which are in turn transformed to a scale of 0-100. Higher scores indicating higher patient satisfaction with medication.
Mean change from Baseline in SF-BPI over time | From Baseline up to Day 150
  Assess the effect of Inclisiran compared to BPA regarding pain-related quality of life using the Short Form Brief Pain Inventory (SF-BPI).
  The SF-BPI is a self-administered standardized fifteen items questionnaire that assesses how pain interferes with or influences a participant's life. The SF-BPI includes two main scores: a pain severity score and a pain interference score. The pain severity score combines the information of the four items about pain intensity, which are rated from 0, no pain, to 10, pain as bad as you can imagine. To derive the pain severity score the average of the four items will be taken. The pain interference is calculated similarly using the seven items regarding pain interference, which are rated from 0, does not interfere, to 10, completely interferes. The pain interference score will be the average of these seven items. Both scores will be between 0 and 10. Higher scores correspond to a poorer condition of the participant.
Proportion of participants with clinically significant change from Baseline in SF-BPI | At day 150
  Proportion of participants with clinically significant change from Baseline [Minimal clinically important difference of 2 points] in SF-BPI, to assess the effect of Inclisiran compared to BPA regarding pain-related quality of life using the Short Form Brief Pain Inventory (SF-BPI).

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (46):
- Germany (46):
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Stuttgart, Baden-Wurttemberg
  - Novartis Investigative Site, Lichtenfels, Bavaria
  - Novartis Investigative Site, Muehldorf Am Inn, Bavaria
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Sulzbach-Rosenberg, Bavaria
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Göttingen, Lower Saxony
  - Novartis Investigative Site, Essen, North Rhine-Westphalia
  - Novartis Investigative Site, Koeln Nippes, North Rhine-Westphalia
  - Novartis Investigative Site, Löhne, North Rhine-Westphalia
  - Novartis Investigative Site, Kaiserslautern, Rhineland-Palatinate
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Leipzig, Saxony
  - Novartis Investigative Site, Jena, Thuringia
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Bad Homburg
  - Novartis Investigative Site, Bad Krozingen
  - Novartis Investigative Site, Bad Oeynhausen
  - Novartis Investigative Site, Bamberg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bremen
  - Novartis Investigative Site, Dessau
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Erfurt
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Falkensee
  - Novartis Investigative Site, Gladbeck
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hoyerswerda
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Ludwigshafen
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Markkleeberg
  - Novartis Investigative Site, Meissen
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Offenbach
  - Novartis Investigative Site, Papenburg
  - Novartis Investigative Site, Pirna
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Rüdersdorf
  - Novartis Investigative Site, Saint Ingbert Oberw
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Völklingen

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com